CLINICAL TRIAL: NCT05381051
Title: Faster Peritoneal Solute Transfer Rate and Survival in a Pre-APD and Icodextrin Peritoneal Dialysis Cohort
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016[099]K
Record Dates: First submitted 2022-05-18; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- original cohort: In the original cohort, 314 patients had catheter implantation between 1st Jan, 2005 to 31st Dec 2009. 269 patients started PD and followed up in our center. 26 patients were excluded due to missing baseline peritoneal membrane function data. 243 patients (n=243, age 53.2±16.3 year) entered the analysis.
- validation cohort: The validation cohort started PD from 2015 to 2018. It was originally designed for a 12 month observational study around fluid balance. 187 patients were in the validation cohort (age 53.0±15.9 year).

SUMMARY:
A fast peritoneal solute transfer rate (PSTR) has been linked to worse survival especially in continuous ambulatory peritoneal dialysis (PD) cohort. In more recent cohorts, where automated PD and icodextrin were more widely used, this association disappears. The current study intended to clarify whether fast PSTR is related to worse outcome in this single center cohort with minimal use of APD and no icodextrin and otherwise modern management practice. Our study found that baseline PSTR predicted patient outcome in univariate survival analysis but not in multivariate analysis. The relationship between comorbidity and faster baseline PSTR may partly explain it.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are Han Chinese;
2. Patients prepare for dialysis in our center, and start PD within 3 months after abdominal catheterization;
3. Patients successfully complete the first peritoneal equilibration test(PET);
4. Follow up regularly in our PD center.

Exclusion Criteria:

1. Patients from hemodialysis to peritoneal dialysis;
2. Patients who need peritoneal dialysis due to transplant-renal loss;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both gender, end stage renal disease on PD treatment
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The relationship between fast PSTR and worse outcome in PD. | The data collection time period of the study is over 10 years.
  Baseline PSTR predicted patient outcome in univariate survival analysis but not in multivariate analysis. The relationship between comorbidity and faster baseline PSTR may partly explain it.